CLINICAL TRIAL: NCT03812185
Title: TEE Image Quality Improvement With Our Devised Transesophageal Echocardiography Probe Cover and Its Effect on Surgical Decision Making
Brief Title: TEE Image Quality Improvement With Our Devised Probe Cover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Henry Ford Hospital (Other)
Responsible Party: Principal Investigator, Yoshihisa Morita, Principal INvestigator, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11958
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Image Quality

STUDY DESIGN:
Intervention Model Description: For intraoperative TEE used cardiac or transplant cases, investigators will compare TEE image quality before and after suctioning using orogastric tube attached TEE probe cover
Masking Description: Since this is a single group study, participant, care provider, and investigator will NOT be masked. However, outcome assessor (who assess image quality and perform measurement using stored TEE images) will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TEE image before and after suctioning orogastric tube (Other): for intraoperative TEE used cardiac or transplant cases, TEE images will be stored before and after suctioning orogastric tube which is attached to TEE probe cover. This Arm is TEE image BEFORE suctioning.
  Interventions: Device: Suctioning orogastric tube which is attached to TEE probe cover

INTERVENTIONS:
Device: Suctioning orogastric tube which is attached to TEE probe cover — Suctioning orogastric tube which is atttached to TEE probe cover.

SUMMARY:
With using suction tube attached TEE probe cover, we will assess its pinpoint suction capacity on image quality and surgical decision making.

DETAILED DESCRIPTION:
Background: Transesophageal echocardiography (TEE) has become a standard intraoperative diagnosis technique for clinical management of patients during cardiac and non-cardiac surgery. Accurate intraoperative diagnosis by TEE improves as image quality improves. Although we recently reported enhanced image quality using a TEE probe with an attached orogastric tube, its clinical significance is still unknown. Also, we are concerned about potential clinical complications including damage to the upper gastrointestinal tract due to its rough surface. Therefore, we devised a new TEE probe cover equipped with a suction catheter and ultrasound gel containing pad that functions as a cushion for preventing surrounding tissue trauma. Our long-term goal is to improve TEE image quality, which will help surgical decision-making with precise assessment. The study population will be elective cardiac cases and liver transplant cases at Henry Ford Hospital. The objective of this grant is to assess the image quality change with our newly designed TEE probe, and its clinical utility on patient care in different types of procedures.

Aim 1. To assess TEE image quality before and after pin-point suctioning with our newly designed TEE probe. We hypothesize that decreasing stomach air between the TEE probe transducer and tissue wall by pin-point suction with our newly designed TEE probe will reduce ultrasound reflection and lead to better image quality.

Aim 2. To evaluate the clinical utility of our newly designed TEE probe cover. We hypothesize our newly designed TEE probe cover will facilitate decision-making for both anesthesiologists and surgeons and it will not increase the occurrence of TEE probe related trauma.

ELIGIBILITY:
Inclusion Criteria: Cardiac procedures and liver transplants which had intraoperative TEE -

Exclusion Criteria: general contraindication with TEE, apparent complications which are related to TEE.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HFHS, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 patients excluded due to resistance to orogastric tube advancement.
Groups:
- TEE Image Before and After Suctioning Orogastric Tube: for intraoperative TEE used cardiac or transplant cases, TEE images will be stored before and after suctioning orogastric tube which is attached to TEE probe cover.
Period: TEE Imaging Before Suctioning
Arm/Group | TEE Image Before and After Suctioning Orogastric Tube
Started | 53
Completed | 50
Not Completed | 3
Not completed — Physician Decision | 3
Period: TEE Imaging After Suctioning
Arm/Group | TEE Image Before and After Suctioning Orogastric Tube
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TEE Image Before and After Suctioning Orogastric Tube
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Age, Continuous [Least Squares Mean (Inter-Quartile Range); unit: years] | 61 [48 to 68]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  gender not known | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Image Quality Assessment Method#1: Difference in Likert Scale Before/After Suctioning
Description: Difference in image quality assessment by Likert scale before/after suctioning, by assessing quality of images stored before/after suctioning. Investigators categorized the quality of all acquired images on a numeric scale (the higher number means higher image quality) based on each investigator's impression (1: very poor, 2: poor, 3: acceptable, 4: good, and 5: very good). Image quality improvement was determined by increased number. Three investigators (A, B, C) assessed the quality of all TEE image sets (i.e. before and after suctioning) post hoc. The acquired numeric scales were combined, and compared before and after suctioning, and calculated how much percentage of patients had improved image quality (i.e. increase in numeric scale), same quality (i.e. same numeric scale), and worsened image quality (i.e. decrease in numeric scale)
Time Frame: TEE image sets were acquired after general anesthesia induction (before suctioning) and after 10minutes (after suctioning), and the outcome was the difference in image quality. In 6-8 months, investigator C did the same analysis on the same images.
Measure: Count of Units; unit: images
Units Other Than Participants: images
Arm/Group | TEE Image Before and After Suctioning Orogastric Tube
Number analyzed (Participants) | 50
Number analyzed (images) | 150
images
  Improved after suction | 83
  Same after suction | 65
  Worse after suction | 2

2. Secondary Outcome: Reproducibility of the LV FAC (Inter-observer)
Description: The reproducibility of the LV FAC was assessed, assuming that better image quality would yield better LV FAC reproducibility. Three investigators (A, B, and C) assessed the quality of all TEE image sets (i.e. before and after suctioning) post hoc. These image sets are combined and assessment was done for each group (i.e. before and after suctioning)
Time Frame: Images were acquired after general anesthesia induction (before suctioning) and after 10minutes (after suctioning images).
Population: Inter-observer intraclass correlation coefficients of LV FAC before and after suctioning.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Units Other Than Participants: Images
Arm/Group | TEE Image Before and After Suctioning Orogastric Tube
Number analyzed (Participants) | 50
Number analyzed (Images) | 150
correlation coefficient
  Intraclass correlation coefficients of LV FAC before suctioning | 0.94 [0.91 to 0.96]
  Intraclass correlation coefficients of LV FAC after suctioning | 0.99 [0.98 to 0.99]

3. Secondary Outcome: Reproducibility of the LV FAC (Intra-observer)
Description: Investigator C analyzed all image sets again in 6-8 months to determine if there was intra-observer variability with the initial assessment of image quality. All investigators were blinded to which images were obtained before or after suctioning.
Time Frame: 6-8 months after initial images obtained during surgery.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Units Other Than Participants: images
Groups:
- Difference in TEE Imaging Before/After Suctioning at 6 Months After the Surgery: Difference in TEE Imaging before/after suctioning at 6 months after the surgery, based on assessor C, to check if there is intraobserver variability.
Arm/Group | Difference in TEE Imaging Before/After Suctioning at 6 Months After the Surgery
Number analyzed (Participants) | 50
Number analyzed (images) | 50
correlation coefficient
  Intraclass correlation coefficients of LV FAC before suctioning | 0.95 [0.91 to 0.99]
  Intraclass correlation coefficients of LV FAC after suctioning | 1.00 [0.99 to 1.00]

4. Secondary Outcome: Reproducibility of the RV FAC (Inter-observer)
Description: The reproducibility of the RV FAC was assessed, assuming that better image quality would yield better RV FAC reproducibility. Three investigators (A, B, and C) assessed the quality of all TEE image sets (i.e. before and after suctioning) post hoc.
Time Frame: Images were acquired after general anesthesia induction (before suctioning) and after 10minutes (after suctioning).
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Units Other Than Participants: Images
Arm/Group | Difference in TEE Imaging Before/After Suctioning at 6 Months After the Surgery
Number analyzed (Participants) | 50
Number analyzed (Images) | 150
correlation coefficient
  Intraclass correlation coefficients of RV FAC before suctioning | 0.89 [0.84 to 0.92]
  Intraclass correlation coefficients of RV FAC after suctioning | 0.90 [0.86 to 0.94]

5. Secondary Outcome: Reproducibility of the RV FAC (Intra-observer)
Description: as for outcome 3
Time Frame: 6-8 months after initial images obtained during surgery.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Units Other Than Participants: Images
Arm/Group | Difference in TEE Imaging Before/After Suctioning at 6 Months After the Surgery
Number analyzed (Participants) | 50
Number analyzed (Images) | 50
correlation coefficient
  Intraclass correlation coefficients of RV FAC before suctioning | 0.88 [0.81 to 0.92]
  Intraclass correlation coefficients of RV FAC after suctioning | 0.85 [0.84 to 0.9]

ADVERSE EVENTS:
Time Frame: 1month
Description: postoperative severe sore throat, dysphagia, bloody aspirate from the OG tube
Groups:
- TEE Image Before Suctioning Orogastric Tube: for intraoperative TEE used cardiac or transplant cases, TEE images will be stored before suctioning orogastric tube which is attached to TEE probe cover.
- TEE Image After Suctioning Orogastric Tube: for intraoperative TEE used cardiac or transplant cases, TEE images will be stored after suctioning orogastric tube which is attached to TEE probe cover.
Arm/Group | TEE Image Before Suctioning Orogastric Tube | TEE Image After Suctioning Orogastric Tube
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT03812185/Prot_SAP_004.pdf
  • Informed Consent Form (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT03812185/ICF_002.pdf